CLINICAL TRIAL: NCT05636176
Title: Effects of Ziltivekimab Versus Placebo on Morbidity and Mortality in Patients With Heart Failure With Mildly Reduced or Preserved Ejection Fraction and Systemic Inflammation
Brief Title: A Research Study to Look at How Ziltivekimab Works Compared to Placebo in People With Heart Failure and Inflammation
Acronym: HERMES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX6018-4915; U1111-1280-0810 (Other: World Health Organization (WHO)); 2022-501939-16-00 (Other: European Medicines Agency (EMA)); jRCT2031230085 (Registry Identifier: jRCT (Japan))
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — ziltivekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ziltivekimab (Experimental): Participants will receive ziltivekimab subcutaneous (s.c.) injection once-monthly and added standard of care for up to 4 years.
  Interventions: Drug: Ziltivekimab
- Placebo (Placebo Comparator): Participants will receive ziltivekimab placebo s.c. injection once-monthly and added standard of care for up to 4 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziltivekimab — Ziltivekimab subcutaneous (s.c.) injection in a pre-filled syringe or a pen-injector once-monthly for up to 4 years.
  Arms: Ziltivekimab
Drug: Placebo — Ziltivekimab placebo s.c. injection in a pre-filled syringe or a pen-injector once-monthly for up to 4 years.
  Arms: Placebo

SUMMARY:
This study will be done to see if ziltivekimab can be used to treat people living with heart failure and inflammation. Participants will either get ziltivekimab or placebo. Participants will get study medicine for once-monthly injections either in a pre-filled syringe to inject the study medicine into a skinfold or a pen-injector to inject the study medicine into flat skin. The study is expected to last for up to 4 years. Participants will have up to 20 clinic visits. Participants will have to use a study app on their phone to record and share information about all their injections of study medicine and to fill in questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Serum high-sensitivity C-reactive protein (hs-CRP) greater than equal to 2 milligrams per liter (mg/L) at screening (visit 1) Disease specific - cardiovascular
* At least one of the following:

  1. N-terminal-pro-brain natriuretic peptide (NT-proBNP) greater than equal to 300 picograms per milliliter (pg/mL) at screening (Visit 1) for patients without ongoing atrial fibrillation/flutter. If ongoing atrial fibrillation/flutter at screening (visit 1), NTproBNP must be greater than equal to 600 pg/mL. Note that the screening electrocardiogram (ECG) must be obtained the same day as sampling for NT-proBNP.
  2. Hospitalisation or urgent/unplanned visit with a primary diagnosis of decompensated heart failure which required intravenous loop diuretic treatment, within the last 9 months prior to screening (visit 1) in combination with NT-proBNP greater than equal to 200 pg/mL at screening (Visit 1) for patients without ongoing atrial fibrillation/flutter. If ongoing atrial fibrillation/flutter at screening (visit 1), NT-proBNP must be greater than equal to 600 pg/mL.
* Diagnosis of heart failure (New York Heart Association [classification] [NYHA] Class II-IV).
* Left ventricular ejection fraction (LVEF) greater than 40 percentage (%) documented by echocardiography within 12 months prior to or at screening (visit 1). The LVEF must be documented in medical records and the most recent measurement must be used to determine eligibility with no interim event signalling potential deterioration in ejection fraction (e.g., myocardial infarction [MI] or heart failure [HF] hospitalisation).
* Structural heart disease and/or functional heart disease documented by echocardiography within 12 months prior to or at screening (visit 1) showing at least one of the following:
* Left atrial (LA) volume index greater than 34 milliliter per meter square (mL/m^2).
* LA diameter greater than equal to 3.8 centimeter (cm).
* LA length greater than equal to 5.0 cm.
* LA area greater than equal to 20 cm square.
* LA volume greater than equal to 55 milliters (mL).
* Intraventricular septal thickness greater than equal to 1.1 cm.
* Posterior wall thickness greater than equal to 1.1 cm.
* Left ventricular (LV) mass index greater than equal to 115 grams per meter square (g⁄m^2 ) in men or greater than equal to 95 g⁄m^2 in women.
* E/e' (mean septal and lateral) greater than equal to 10.
* e' (mean septal and lateral) less than 9 centimeter per second (cm/s).
* No heart failure hospitalisations or urgent heart failure visits between screening (visit 1) and randomisation (visit 2).

Exclusion Criteria:

Medical conditions - cardiovascular

* Myocardial infarction, stroke, unstable angina pectoris, transient ischaemic attack, or heart failure hospitalisation, within 30 days prior to screening (visit 1).
* Systolic blood pressure greater than equal to 180 millimeters of mercury (mmHg) at screening (visit 1). If the systolic blood pressure is 160-179 mmHg, the patient should be receiving greater than equal to 3 antihypertensive drugs. (Note: Potential participants may be retested for this criterion within the visit window and without rescreening, at the discretion of the investigator).
* Heart rate above 110 or below 40 beats per minute as evaluated on the electrocardiogram (ECG) performed at screening (visit 1) (Note: Potential participants may be retested for this criterion within the visit window and without rescreening, at the discretion of the investigator).
* Planned coronary, carotid or peripheral artery revascularisation known during the screening period (visit 1). (Note: Planned coronary angiogram is not exclusionary).
* Planned cardiac device or atrial flutter/atrial fibrillation ablation procedure known during the screening period (visit 1).
* Major cardiac surgical, non-cardiac surgical, or major endoscopic procedure (thoracoscopic or laparoscopic) within the past 60 days prior to randomisation (visit 2) or any major surgical procedure planned at the time of randomisation (visit 2).
* Heart failure due to infiltrative cardiomyopathy (e.g., sarcoid, amyloid), arrhythmogenic right ventricular cardiomyopathy, Takutsubo cardiomyopathy, genetic hypertrophic cardiomyopathy or obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, cardiac tamponade, uncorrected more than moderate primary valve disease.
* Primary pulmonary hypertension, chronic pulmonary embolism, severe pulmonary disease including COPD.
* Any other condition judged by the investigator that could account for heart failure symptoms and signs (e.g., anaemia, hypothyroidism).

Medical conditions - infections/immunosuppression

- Clinical evidence of, or suspicion of, active infection at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5600 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2027-07-02 (Estimated); Study Completion 2027-07-02 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of a Composite Heart Failure Endpoint Consisting of: Cardiovascular (CV) Death, Heart Failure (HF) Hospitalisation or Urgent HF Visit | From randomisation (month 0) to end of study (up to 48 months)
  Measured in months.

SECONDARY OUTCOMES:
Time to First Occurrence of 4-point Expanded Composite HF Endpoint, a Composite Endpoint Consisting of: CV Death, HF Hospitalisation or Urgent HF Visit, Non-fatal Myocardial Infarction (MI), Non-fatal Stroke | From randomisation (month 0) to end of study (up to 48 months)
  Measured in months.
Number of CV Deaths, HF Hospitalisations or Urgent HF Visits (First and Recurrent) | From randomisation (month 0) to end of study (up to 48 months)
  Measured as count of event.
Time to Occurrence of CV Death | From randomisation (month 0) to end of study (up to 48 months)
  Measured in months.
Time to Occurrence of all-cause Death | From randomisation (month 0) to end of study (up to 48 months)
  Measured in months.
Time to First Occurrence of 4-point Expanded Composite HF Endpoint, a Composite Endpoint Consisting of: All-cause Death, HF Hospitalisation or Urgent HF Visit, Non-fatal MI, Non-fatal stroke | From randomisation (month 0) to end of study (up to 48 months)
  Measured in months.
Hierarchical Composite of: Time to All-cause Death, Number of HF Hospitalisations or Urgent HF Visits, Time to First HF Hospitalisation or Urgent HF Visit, difference of at least 5 in KCCQ clinical summary score change from baseline to 12 months | From randomisation (month 0) to end of study (up to 48 months)
  Kansas City Cardiomyopathy Questionnaire (KCCQ) measures Health-Related Quality of Life (HRQOL) and is a disease-specific health status instrument for HF. Score ranges from 0 to 100, with 0 as the lowest score and 100 as the highest score. Higher scores indicate better health status, fewer symptoms, and greater disease-specific health related quality of life, respectively. Measured as total wins for each treatment group.
Time to First Occurrence of HF Hospitalisation or Urgent HF Visit | From randomisation (month 0) to end of study (up to 48 months)
  Measured in months.
Number of Events of Atrial Fibrillation | From randomisation (month 0) to end of study (up to 48 months)
  Measured as count of event.
Change in KCCQ Clinical Summary Score | From randomisation (month 0) to 12 months
  KCCQ measures Health-Related Quality of Life (HRQOL) and is a disease-specific health status instrument for HF. Score ranges from 0 to 100, with 0 as the lowest score and 100 as the highest score. Higher scores indicate better health status, fewer symptoms, and greater disease-specific health related quality of life, respectively. Measured as score.
Improvement of 5 Points or More in KCCQ Clinical Summary Score (Yes/No) | From randomisation (month 0) to 12 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ) measures Health-Related Quality of Life (HRQOL) and is a disease-specific health status instrument for HF. Score ranges from 0 to 100, with 0 as the lowest score and 100 as the highest score. Higher scores indicate better health status, fewer symptoms, and greater disease-specific health related quality of life, respectively. Measured as count of participant.
Improvement of 10 Points or More in KCCQ Clinical Summary Score (Yes/No) | From randomisation (month 0) to 12 months
  Kansas City Cardiomyopathy Questionnaire (KCCQ) measures Health-Related Quality of Life (HRQOL) and is a disease-specific health status instrument for HF. Score ranges from 0 to 100, with 0 as the lowest score and 100 as the highest score. Higher scores indicate better health status, fewer symptoms, and greater disease-specific health related quality of life, respectively. Measured as count of participant.
Improvement in New York Heart Association (Classification) [NYHA Class] (Yes/No) | From randomisation (month 0) to 12 months
  NEW YORK HEART ASSOCIATION CLASSIFICATION (NYHA) Class I: Participant with cardiac disease but without resulting limitations of physical activity.
  Class II: Participants with cardiac disease resulting in slight limitation of physical activity.
  Class III: Participants with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Participants with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Measured as count of participant.
Time to First Occurrence of a Composite Chronic Kidney Disease (CKD) Endpoint Consisting of: CV death, Onset of Persistent Greater Than Equal To 40 Percentage Reduction in eGFR (CKD- EPI) compared with baseline; Kidney failure | From randomisation (month 0) to end of study (up to 48 months)
  eGFR = estimated glomerular filtration rate; CKD-EPI = chronic kidney disease - epidemiology collaboration. Kidney failure defined as: death from kidney failure, onset of persistent eGFR less than 15 milliliters per minute (mL/min)/1.73 meter square (m^2) (CKD-EPI), initiation of chronic kidney replacement therapy (maintenance dialysis or kidney transplantation). Measured in months.
Change in Estimated Glomerular Filtration Rate (eGFR) (Chronic Kidney Disease - Epidemiology Collaboration [CKD-EPI]) | From randomisation (month 0) to 12 months
  Measured as mL/min/1.73 m^2.
Annual Rate of Change in eGFR (CKD-EPI) (Total eGFR Slope) | From randomisation (month 0) to end of study (up to 48 months)
  Measured as mL/min/1.73 m^2/year.
Number of Hospitalisations With Infection as Primary Cause or Death Due to Infection | From randomisation (month 0) to end of study (up to 48 months)
  Measured as count of event.
Change in High-sensitivity C-reactive Protein (hs-CRP) | From randomisation (month 0) to 12 months
  Measured as ratio to baseline.
Change in N-terminal-pro-brain Natriuretic Peptide (NT-proBNP) | From randomisation (month 0) to 12 months
  Measured as ratio to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (991):
- United States (167):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - Eastern Shore Rsrch Inst, LLC, Fairhope, Alabama
  - Heart Center Rsrch_Hunstville, Huntsville, Alabama
  - Banner University Medical Ctr, Phoenix, Arizona
  - Cardiology & Medicine Clinic, Little Rock, Arkansas
  - InvivoCure -2, Alhambra, California
  - National Heart Institute Cal, Beverly Hills, California
  - Valley Clinical Trials, Covina, California
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Purushotham & Akther Kotha MD, inc., La Mesa, California
  - VA Loma Linda Hlthcr Sys, Loma Linda, California
  - Biopharma Clinical Research Services, LLC, Los Angeles, California
  - VA Greater Los Angeles Hlthcare System, Los Angeles, California
  - VAGrtrLosAngelesHlthcareSystem, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - UCI Health, Orange, California
  - Stanford Univ School of Med, Palo Alto, California
  - San Diego Cardiac Center, San Diego, California
  - North America Research Institute, San Dimas, California
  - Manshadi Heart Institute, Stockton, California
  - Lundquist Inst-Biomed Innovtn, Torrance, California
  - InvivoCure, Van Nuys, California
  - Rocky Mountain Regional VAMC, Aurora, Colorado
  - InvivoCure -2, Denver, Colorado
  - S Denver Cardiology Associates, Littleton, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Cardiology Associates of Fairfield County, Stamford, Connecticut
  - Pioneer Clinical Studies-Coral Gables, Coral Gables, Florida
  - Nature Coast Clin Rsrch_Crystal River, Crystal River, Florida
  - Integrative Research Assoc Inc, Fort Lauderdale, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - Memorial Region Hosp_Hollywood, Hollywood, Florida
  - E Coast Inst for Rsrch LLC_Jacksonville, Jacksonville, Florida
  - Jacksonville Ctr for Clin Res, Jacksonville, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - Baptist Health South Florida, Miami, Florida
  - NCH Research Institute, Naples, Florida
  - Amavita Research Services, LLC, North Miami Beach, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - St Johns Ctr Clin Rsch-St. Aug, Saint Augustine, Florida
  - Cardio Partners Clin Res Inst, Wellington, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Guardian Research Org LLC, Winter Park, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Emory University School of Medicine_Atlanta, Atlanta, Georgia
  - NSC Research, Inc, Johns Creek, Georgia
  - GA Arrhythmia Cons & Rsch Inst, Macon, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - St. Luke's Idaho Cardiology Associates, Meridian, Idaho
  - Endeavor Health Clinical Operations-NCH, Arlington Heights, Illinois
  - Advocate Good Samaritan, Downers Grove, Illinois
  - Chicago Medical Research LLC, Hazel Crest, Illinois
  - Midwest Cardiovascular Institute, Naperville, Illinois
  - OSF HealthCare_Cardiovasc Inst, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Midwest Cardiovascu Rsrch Foundation, Elkhart, Indiana
  - Asha Clinical Rsch-Munster, LLC, Hammond, Indiana
  - Franciscan Network-IN Heart PHY, Indianapolis, Indiana
  - Witham Health Services, Lebanon, Indiana
  - Cardiovascular Rsrch of NW_IN, Munster, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - University Of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Midwest Heart & Vasc Spec, Overland Park, Kansas
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - The Research Group of Lexington LLC, Lexington, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - LOUISIANA HEART Center, Bogalusa, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ascension Saint Agnes Heart Ca, Baltimore, Maryland
  - Johns Hopkins University_Baltimore, Baltimore, Maryland
  - Capitol Cardiology Assoc_Lanham, Lanham, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - University of Michigan Medicine, Ann Arbor, Michigan
  - Detroit Med Center-Wayne State, Detroit, Michigan
  - Henry Ford Hlth System_Detroit, Detroit, Michigan
  - Elite Research Center, Flint, Michigan
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - Trinity Health Michigan Heart, Ypsilanti, Michigan
  - Fairview Health Services, Maplewood, Minnesota
  - Minneapolis VA Health Care Sys, Minneapolis, Minnesota
  - Hawthorne Health, Diamondhead, Mississippi
  - Cardiolg Assoc Rsch LLC_Tupelo, Tupelo, Mississippi
  - St Louis Heart & Vascular, P.C., St Louis, Missouri
  - Logan Health Research, Kalispell, Montana
  - Univ. of Nebraska Medical Center_Omaha, Omaha, Nebraska
  - Palm Research Center Inc., Las Vegas, Nevada
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Heart House_Elmer, Elmer, New Jersey
  - NJ Heart, Linden, New Jersey
  - Barnabas Health, Livingston, New Jersey
  - Inspira Health, Mullica Hill, New Jersey
  - Saint Michael's Med Ctr NJ, Newark, New Jersey
  - The Valley Hosptial, Ridgewood, New Jersey
  - Capital Cardiology Associates_Albany, Albany, New York
  - University at Buffalo_Erie County Med Ctr, Buffalo, New York
  - Marian David, MD, PC, Kew Gardens, New York
  - Mount Sinai Hosp at NYC, New York, New York
  - NY Presbyt Hosp-W Cornell Med, New York, New York
  - Harlem Cardiology_Madison ave, New York, New York
  - Laurelton Heart Specialist PC, Rosedale, New York
  - Saratoga Clinical Research, Saratoga Springs, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Chear Center LLC, The Bronx, New York
  - UNC Cardiology Outpatient Ctr, Chapel Hill, North Carolina
  - Hawthorne Health NC, Concord, North Carolina
  - Duke University, Durham, North Carolina
  - Medication Mgmnt, LLC_Grnsboro, Greensboro, North Carolina
  - Duke University/Southeastern, Lumberton, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Aultman Hospital, Canton, Ohio
  - K&R Research Llc, Marion, Ohio
  - Rama Research LLC, Marion, Ohio
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Capital Area Research LLC, Camp Hill, Pennsylvania
  - Penn State Hlth Holy Spirit Med Ctr, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Heart Grp_ Lancaster Gen Hlth, Lancaster, Pennsylvania
  - Thomas Jefferson University_Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Penn State Health-Berks Cardiology, Wyomissing, Pennsylvania
  - Prisma Health-Midlands, Columbia, South Carolina
  - Monument Health Clinical Rsrch, Rapid City, South Dakota
  - Sanford Health_Sioux Falls, Sioux Falls, South Dakota
  - Apex Research Foundation, LLC, Jackson, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Tennova HC Turkey Creek MC, Knoxville, Tennessee
  - Heart MD_Allen TX, Allen, Texas
  - PharmaTex Research, LLC, Amarillo, Texas
  - Austin Heart, Austin, Texas
  - UTD SW Medical Center-Dallas, Dallas, Texas
  - Dallas Heart and Vascular, Duncanville, Texas
  - David Turbay, MD, PLLC, El Paso, Texas
  - Biopharma Informatic_Houston, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Texas Heart Inst Medical Ctr, Houston, Texas
  - UT Physicians - Houston Medical Center, Houston, Texas
  - Card Specialists of Willowbrook, Houston, Texas
  - Texas Institute of Cardiology PA, McKinney, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - Audie L. Murphy VA Hospital, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - James River Cardiology, Chesterfield, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - Sentara Health Research Center, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
  - VA Medical Center_Salem, Salem, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Valley Health Link, Winchester, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center_Seattle, Seattle, Washington
  - Providence Med Research Ctr, Spokane, Washington
  - WVU Heart & Vascular Institute, Morgantown, West Virginia
  - William S Middleton Mem VA Hosp, Madison, Wisconsin
  - Aurora St. Luke's Medi Ctr, Milwaukee, Wisconsin
- Argentina (19):
  - Mautalen Salud e investigación, CABA, Buenos Aires
  - CEMEDIC, CABA, Buenos Aires
  - Centro de Investigaciones Médicas Clínica de Fracturas y Or, Mar del Plata, Buenos Aires
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata, Buenos Aires
  - Fundacion Favaloro, CABA, Buenos Aires, Argentina
  - Centro de Investigaciones Clinica Baigorria, Granadero Baigorria, Santa Fe Province
  - Centro de Investigaciones Clinica Baigorria, Santa Fé, Santa Fe Province
  - DIM Clinica Privada, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Fundacion Favaloro, CABA
  - CEMEDIC, CABA
  - Instituto de Cardiología de Corrientes, Corrientes
  - Instituto de Investigaciones Clinicas Mar Del Plata, Mar del Plata
  - Instituto de Investigaciones Clinicas, Mar del Plata
  - Centro de Investigaciones Médicas Clínica de Fracturas y Or, Mar del Plata
  - Instituto de Investigaciones Clinicas San Nicolás, San Nicolás
  - Centro de investigaciones Clinicas del Litoral, Santa Fe
  - CEDIR - Centro de diagnóstico y rehabilitación Santa Fe, Santa Fe
- Australia (17):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repatriation General Hospital - Cardiology Department, Concord, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Sydney Cardiometabolic Centre, Liverpool, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Heart of Australia, Chelmer, Queensland
  - Townsville University Hospital, Douglas, Queensland
  - Nightingale Research, Adelaide, South Australia
  - Royal Adelaide Hospital Cardiovascular Clinical Trials, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Frankston Hospital, Frankston, Victoria
  - Adrian Costa Clinical Trials Centre, Geelong, Victoria
  - Barwon Health (The Geelong Hospital), Geelong, Victoria
  - HeartWest Cardiology - Hoppers Crossing, Hoppers Crossing, Victoria
  - Epworth HealthCare, Richmond, Victoria
  - Clinitrials, Perth, Western Australia
- Austria (8):
  - Krankenhaus St. Josef Braunau, Braunau am Inn
  - Medizinische Universität Graz, Graz
  - Fließer-Görzer [Ordination], Saint Stefan
  - Uniklinikum Salzburg Kardiologie, Salzburg
  - Medizinische Universität Wien, Vienna
  - Klinik Favoriten, Vienna
  - Klinik Ottakring, Vienna
  - Imed 19- privat, Vienna
- Belgium (6):
  - AZORG Aalst - Moorselbaan, Aalst
  - UZ Brussel, Brussels
  - UZA - UZ Antwerpen - Cardiology Department, Edegem
  - Ziekenhuis Oost-Limburg AV - Cardiology, Genk
  - AZ Groeninge - Kortrijk - Cardiology, Kortrijk
  - CHR de la Citadelle, Liège
- Bosnia and Herzegovina (3):
  - University Clinical Centre of the Republic Srpska, Banja Luka
  - Dr. Abdulah Nakas General Hospital, Sarajevo
  - University Clinical Centre Sarajevo, Sarajevo
- Brazil (23):
  - Centro de Diag. e Pesquisa da Osteoporose do Espírito Santo, Vitória, Espírito Santo
  - CCIH-Consultoria em Controle de Infecção Hospitalar Ltda, Belo Horizonte, Minas Gerais
  - NUPEC Cardio, Belo Horizonte, Minas Gerais
  - Eurolatino Medical Research Center, Uberlândia, Minas Gerais
  - Sociedade Hospitalar Angelina Caron, Brazil, Campina Grande do Sul, Paraná
  - PUCPR - Pontificia Universidade Catolica do Parana, Curitiba, Paraná
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Associação Lar São Francisco de Assis na Providência de Deus - Bragança Paulista, Bragança Paulista, São Paulo
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - PUCCAMP - Hospital e Maternidade Celso Pierro, Campinas, São Paulo
  - i9 Pesquisas Clínicas, Campinas, São Paulo
  - Unidade de Pesquisa Clínica do Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - CIP Centro Integrado de Pesquisas do Hospital de Base, São José do Rio Preto, São Paulo
  - Instituto de Moléstias Cardiovasculares de Tatuí Ltda, Tatuí, São Paulo
  - Integral Pesquisa e Ensino, Votuporanga, São Paulo
  - Jmf Clínica Do Coração Ltda, Aracaju
  - Hospital de Clínicas da Universidade Federal de Goiânia, Goiânia/GO
  - ICM - Instituto do Coração de Marília, Marília/SP
  - Hospital Mãe de Deus - Porto Alegre, Porto Alegre/RS
  - PROCAPE, Recife/PE
  - Hospital São Lucas Copacabana, Rio de Janeiro
  - Instituto D'or de Pesquisa e Ensino, Rio de Janeiro
  - Universidade Federal de São Paulo - UNIFESP, São Paulo/SP
- Bulgaria (29):
  - MHAT Heart and Brain EAD, Burgas
  - Medical Centre - Avitsena EOOD, Kardzhali
  - Medical centre "Zdrave 1" OOD, Kozloduy
  - Medical centre Zdrave 1 OOD, Kozloduy
  - Medical Centre Hera - Kyustendil EOOD, Kyustendil
  - DCC 1 - Lom EOOD, Lom
  - Diagnostic Consulting Center 1- Lom EOOD, Lom
  - "MHAT - UniHospital" OOD, Panagyurishte
  - MHAT - UniHospital OOD, Panagyurishte
  - Medical center Medconsult Pleven OOD, Pleven
  - UMHAT "Dr. Georgi Stranski" Pleven, Pleven
  - MHAT Heart and Brain, Pleven
  - UMHAT - Plovdiv AD, Plovdiv
  - UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Cardiology, Plovdiv
  - MHAT Sveta Karidad EAD, Plovdiv
  - MC Health Care OOD, Sandanski, Sandanski
  - 'Medical Center Hipokrena' EOOD, Sevlievo
  - Medical Center Hipokrena EOOD, Sevlievo
  - Medical Centre Cardiomed 2020 EOOD, Sliven
  - DCC Ascendent OOD, Sofia
  - MHAT Knyaginya Klementina - Sofia EAD, Sofia
  - NMTH Tsar Boris III, Sofia
  - MHAT Sveta Sofia EOOD, Sofia
  - DCC Aleksandrovska EOOD, Sofia
  - Medical center ISUL - Tsaritsa Yoanna EOOD, Sofia
  - Medical Centre Intermedica OOD, Sofia
  - Medical center Zara-Med EOOD, Stara Zagora
  - MDHAT Dr. Stephen Cherkezov AD, Veliko Tarnovo
  - MC Nevromedics EOOD, Cardiology, Veliko Tarnovo
- Canada (36):
  - University of Calgary_Calgary, Calgary, Alberta
  - Alta Clinical Research, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - North Shore Heart Centre, North Vancouver, British Columbia
  - SMH Cardiology Clinical Trials Inc., Surrey, British Columbia
  - Ctr for Cardiovascular Innovation, Vancouver, British Columbia
  - St Pauls Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Nova Scotia Health, Halifax, Nova Scotia
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Saul Vizel Pro. Med. Corp, Cambridge, Ontario
  - Health Sciences North Rsrch Inst, Greater Sudbury, Ontario
  - Dawson Clinical Research, Guelph, Ontario
  - Hamilton Hlth Sc. - General Site, Hamilton, Ontario
  - St. Joseph's Hospital, London, Ontario
  - Partnrs Adv Cardio Eval (PACE), Newmarket, Ontario
  - North York Diagn & Cardiac Ctr, North York, Ontario
  - Centricity Research Oshawa, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - St. Michael's Hospital_Toronto, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Clinical Research Solutions Inc., Waterloo, Ontario
  - CPS Research, Waterloo, Ontario
  - Winchester Dist Memorial Hosp, Winchester, Ontario
  - Viacar Recherche Clinique Inc., Longueuil, Quebec
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - CHU de Montréal, Montreal, Quebec
  - CardioVasc HR Inc, Saint-Jean-sur-Richelieu, Quebec
  - CIUSSS de l'E CHUS_Sherbrooke, Sherbrooke, Quebec
  - CISSSL Hôsp Pierre-Le Gardeur, Terrebonne, Quebec
  - Ctr de méd métab de Lanaudière, Terrebonne, Quebec
  - Diex Recherche Trois-Rivieres, Trois-Rivières, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- China (54):
  - The First Hospital of Anhui University of Science & Technology (Huainan First People's Hospital)-Cardiology, Huainan, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences Fuwai Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital-Cardiology, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University-Cardiology, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - The Second Hospital & Clinical Medical School, Lanzhou University-Internal Medicine & Cardiovascular, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen Universtiy, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College-Cardiovascular, Shantou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The First Hospital of Hebei Medical University-Cardiovascular, Shijiazhuang, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University-Cardiovascular, Harbin, Heilongjiang
  - Wuhan Asia Heart Hospital-Department of Cardiovascular, Wuhan, Hubei
  - Renmin Hospital of Wuhan University-Cardiology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Changsha Central Hospital, Changsha, Hunan
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University-Cardiology, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Affiliated Hospital of Nanchang University-Cardiology, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University-Cardiology, Changchun, Jilin
  - Jilin Province People's Hospital-Cardiology, Changchun, Jilin
  - Siping Central People's Hospital-Cardiology, Siping, Jilin
  - The People's Hospital of Liaoning Province-Cardiology, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an JiaoTong University-Cardiovascular, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital-Cardiology, Xi'an, Shaanxi
  - The Affiliated Hospital of Jining Medical University-Cardiology, Jining, Shandong
  - Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University-Cardiology, Shanghai, Shanghai Municipality
  - Mianyang Central Hospital-Cardiology, Mianyang, Sichuan
  - Tianjin Union Medical Center, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Lishui People's Hospital-Cardiology, Lishui, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
  - The First Affiliated Hospital of WMU-Cardiology, Wenzhou, Zhejiang
  - Chongqing University Three Gorges Hospital, Chongqing
  - Shanghai Xuhui Central Hospital, Shanghai
- Colombia (14):
  - Hospital General de Medellin, Medellín, Antioquia
  - Rodrigo Botero S.A.S, Medellín, Antioquia
  - IPS Centro Cientifico Asistencial Jose Luis Accini SAS, Barranquilla, Atlántico
  - Clinica de la Costa, Barranquilla, Atlántico
  - Fundación Hospital Universidad del Norte, Soledad, Barranquilla
  - IPS médicos Internistas de Caldas S.A.S., Manizales, Caldas Department
  - Centro de Atención e Investigación Médica S.A.S. (CAIMED SAS), Chía, Cundinamarca
  - Unidad de Estudios Clínicos de la Fundación Cardiovascular de Colombia, Bucaramanga-piedecuesta, Valle Del Menzuli - Santander, Santander Department
  - Clinica Imbanaco SAS, Cali, Valle del Cauca Department
  - Corazón IPS S.A.S, Barranquilla
  - Fundacion del Caribe para la Investigacion Biomedica-BIOS, Barranquilla
  - Fundación Santa Fe de Bogotá, Bogotá
  - Promotora Medica Las Americas S.A., Medellín
  - CardiovidCentro Cardiovascular Colombiano ClinicaSantaMaria, Medellín
- Croatia (16):
  - Poliklinika Aritmija, Zagreb, City of Zagreb
  - University Hospital Centre Zagreb, Zagreb, City of Zagreb
  - KB Dubrava, Zavod za bolesti srca i krvnih zila, Zagreb, City of Zagreb
  - Poliklinika Solmed, Zagreb, City of Zagreb
  - Specijalna bolnica za medicinsku rehabilitaciju Krapinske Toplice_Cardiology, Krapinske Toplice, Krapinsko Zagorska County
  - Poliklinika Medikol_Cakovec_Cardiology, Čakovec
  - Zupanijska bolnica Cakovec, Čakovec
  - Internacionalni medicinski centar PRIORA, Čepin
  - Opca bolnica Karlovac_Cardiology, Karlovac
  - Opca bolnica Karlovac, Karlovac
  - Klinicki Bolnicki Centar Osijek_Cardiology, Osijek
  - Clinical Hospital Centre Rijeka_Cardiology, Rijeka
  - Specijalna bolnica Medico, Rijeka
  - KBC Split_Cardiology, Split
  - University Hospital Sveti Duh, Zagreb
  - Poliklinika Magnolija d.o.o., Zagreb
- Czechia (16):
  - Kardiologie MUDr. Libor Nechvátal s.r.o., Brno
  - Amkardia s.r.o., Brno
  - FN Hradec Kralove, Hradec Králové
  - KARDIOLOGIE - LIBEREC s.r.o., Liberec
  - Fakultni nemocnice Plzen - Lochotin, Plzen - Lochotín
  - Policska nemocnice, Polička
  - Poličská nemocnice s.r.o., Polička
  - Kardiologická a interní ambulance, Prague
  - Kardiologie Vinohrady s.r.o., Prague
  - Fakultní poliklinika VFN ambulance Srdecniho selhani, Prague
  - Nemocnice Slany Kardiologie, Slaný
  - Nemocnice Slany, Slaný
  - Vseobecna kardiologicka ambulance, Tábor
  - Všeobecná kardiologická ambulance s.r.o., Tábor
  - Kardiologie Trutnov Ferkl, Trutnov
  - Clinical Trials Service s.r.o., Uherské Hradiště
- Denmark (7):
  - Herlev Hospital - Afdeling for Hjertesygdomme, Forskning 1, Herlev, Capital Region
  - Kardiologisk Odense & Svendborg, Svendborg, Region South
  - Svendborg Sygehus - Kardiologisk, Svendborg, Region South
  - Aarhus Universitetshospital, Hjertesygdomme, Aarhus N
  - Aarhus Universitetshospital, Skejby Hjertesygdomme, Aarhus N
  - Bispebjerg og Frederiksberg Hospital, Frederiksberg
  - Sjællands Universitetshospital, Roskilde - Kardiologisk Afdeling, Roskilde
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Finland (6):
  - HUS, Sydän- ja keuhkokeskus, kardiologian tutkimusyksikkö, HUS
  - StudyCor, Jyväskylä
  - Health Step Finland Oy, Kuopio
  - Seinäjoen keskussairaala, Seinäjoki
  - TAYS Sydänsairaala, Tampere
  - TYKS Sydänkeskus, Turku
- France (10):
  - Centre Hospitalier Universitaire Grenoble Alpes-Site Nord Michallon, La Tronche
  - Hôpital Arnaud de Villeneuve_Service de Cardiologie, Montpellier
  - Aphp-Hopital Lariboisiere-1, Paris
  - Aphp-Hopital La Pitie Salpetriere-1, Paris
  - Centre Hospitalier de Pau - Hopital Francois Mitterrand, Pau
  - CENTRE HOSPITALIER UNIVERSITAIRE DE POITIERS - Centre Cardio Vasculaire, Poitiers
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Intercommunal Toulon La Seine-Sur-Mer - Hopital Sainte Musse, Toulon
  - CENTRE HOSPITALIER UNIVERSITAIRE DE TOULOUSE-HOPITAL RANGUEIL_Service de Cardiologie, Toulouse
  - Chru de Nancy - Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (31):
  - Uniklinik Aachen - Med. Klinik I, Aachen
  - Velocity - Clinical Research Germany GmbH, Berlin
  - Charite Universitatsmedizin Berlin KöR, Berlin
  - Charité - Campus Virchow-Klinikum - Kardiologie, Angiologie und Intensivmedizin (CRU), Berlin
  - Uniklinik Klinikum Bielefeld - Kardiologie und Internist. Intensivmedizin, Bielefeld
  - Kath. Klinikum Bochum gGmbH - St. Josef-Hospital Kardiologie, Bochum
  - Kardiologisch-Angiologische Praxis Herzzentrum Bremen, Bremen
  - Kath. St. Paulus GmbH - St Johannes Hospital Dortmund - Kardiologie, Dortmund
  - Facharztzentrum Dresden Betriebsgesellschaft mbH, Dresden
  - Cardiologicum Dresden und Pirna - MVZ "Am Felsenkeller" (Dresden), Dresden
  - Uniklinik TU Dresden - Herzzentrum Dresden GmbH, Dresden
  - Zentrum fuer klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - MVZ CCB Frankfurt und Main-Taunus GbR, Frankfurt
  - Universitätsklinikum Frankfurt aM - Kardiologie, Frankfurt am Main
  - Universitätsklinikum Freiburg - Medical Center, Freiburg im Breisgau
  - Justus-Liebig-Universität Gießen - Kardiologie, Giessen
  - Uni-Med. Göttingen - Kardiologie, Pneumologie, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf - University Medical Center Hamburg-Eppendorf, Hamburg
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Kardiologie Hassloch, Haßloch
  - Universität des Saarlandes - Innere Med. III, Homburg
  - Uniklinik Jena - Kardiologie, Jena
  - Kardiopraxis Schirmer, Kaiserslautern
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für Kardiologie, Leipzig
  - Gesundheitscentrum Mainz (Regner / Schmitt), Mainz
  - zero PRAXEN Mannheim-Schwetzingerstadt, Mannheim
  - LMU Klinikum München Klinik und Poliklinik 1, München
  - Kardiologische Gemeinschaftspraxis Papenburg, Papenburg
  - Herz-Kreislauf-Zentrum Klinikum Hersfeld-Rotenburg GmbH, Rotenburg A.d. Fulda
  - Al-Zoebi, Wermsdorf
  - Universitatsklinikum Würzburg - Zentrum für Herzinsuffizienz, Würzburg
- Greece (26):
  - Alexandra General Hospital, Therapeutic Clinic, Athens, Attica
  - University General Hospital Of Heraklion - Cardiology Department, Heraklion, Crete
  - General Hospital of Athens "Elpis" - Cardiology Department, Ampelokipoi/Athens
  - 'G. Gennimatas' General Hospital of Athens - Cardiology Department, Athens
  - Hippokration Hospital, Athens
  - Thoracic General Hospital Of Athens I Sotiria - Cardiology Department, Athens
  - Konstantopouleio G.H. of Athens, "Agia Olga", Athens
  - "Hygeia" General Hospital of Athens, Athens
  - Iatriko Athinon (Athens Medical Canter), Athens
  - Genl Hospital of Athens Ippokrateio,A' Cardiology Univ dpt, Athens
  - U.G.H of Athens "Attikon", Chaidari, Athens
  - General Hospital of Kalamata - Cardiology Department, Chalcis
  - General Hospital of Chios "Skilitsio" - Cardiology Clinic, Chios
  - General Hospital Venizeleio-Pananeio - Cardiology department, Heraklion
  - Venizeleio Pananeio, Heraklion
  - General Hospital of Kalamata - Cardiology Department, Kalamata
  - General Hospital of Kalamata, Kalamata
  - General Oncological Hospital of Kifissia Agioi Anargyroi - Cardiology Clinic, Kifissia
  - Univ Gen Hospital Larisa, Cardiology Medicine Clinic, Larissa
  - General Hospital Of Mytilene Vostanio - Cardiology Department, Mytilene
  - Geniko Nosokomeio Peiraia Tzaneio - Cardiology department, Piraeus
  - Iatriko Athinon (Athens Medical Canter), Pylea, Thessaloniki
  - General University Hospital of Patras, Rio Patras
  - General Hospital of Thessaloniki 'G. Gennimatas - Cardiology Department, Thessaloniki
  - "AHEPA" University General Hospital of Thessaloniki, Thessaloniki
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
- Hungary (20):
  - PTE ÁOK I. sz. Belgyógyászati Klinika, Pécs, Baranya
  - Dr. Lakatos Ferenc Kardiológus ,Belgyógyász Magán szakrendelés, Békéscsaba, Bekes County
  - Arina Trial Research Kft., Orosháza, Bekes County
  - Lausmed Kft., Baja, Bács-Kiskun county
  - Szegedi Tudományegyetem II. sz Belgyógyászati és Kardiológia, Szeged, Csongrád-Csanád
  - Selye János Kórház, Komárom, Komárom-Esztergom
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County
  - Léda Platán Magánklinika, Zalaegerszeg, Zala County
  - EURÉKA-CENTER Orvosi és Szolgáltató Betéti Társaság, Baja
  - DRC Kft., Balatonfüred
  - Tagore Medical Center, Balatonfüred
  - Betegápoló Irgalmasrend, Budai Irgalmasrendi Kórház, Budapest
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászat, Budapest
  - Észak-Pesti Centrumkórház Honvédkórház, Budapest
  - Jahn Ferenc Dél-pesti Kórház és Rendelőintézet, Budapest
  - Békés Vármegyei Központi Kórház, Gyula
  - Borsod-Abaúj-Zemplén Vármegyei Központi Kórház És Egyetemi Oktatókórház, Miskolc
  - Coromed SMO Kft., Pécs
  - Szegedi Tudományegyetem, Szeged
- India (54):
  - Lalitha Super Specialities Hospital, Guntur, Andhra Pradesh
  - Ramesh Hospitals, Vijayawada, Andhra Pradesh
  - Siddhartha Medical College & Government General Hospital, Vijaywada, Andhra Pradesh
  - GNRC Hospital, Guwahati, Assam
  - Sardar Vallabhbhai Patel Institute of Medical Sciences and Research, Ahmedabad, Gujarat
  - CIMS- Care Institute of Medical Sciences, Ahmedabad, Gujarat
  - EPIC Hospital, Ahmedabad, Gujarat
  - Shri B. D. Mehta Mahavir Heart Institute, Surat, Gujarat
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - Medanta - The Medicity Multi-Speciality Hospital, Gurugram, Gurugram, Haryana
  - Manipal Hospital, Old Airport Road, Bengaluru, Bangalore, Karnataka
  - KLES Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi, Karnataka
  - Sri Jayadeva Institute of Cardiovascular Sciences & Research, Bengaluru, Karnataka
  - Narayana Institute of Cardiac Sciences, Bengaluru, Karnataka
  - Lisie Hospital, Kochi, Kerala
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Government Medical College and Super Speciality Hospital, Nagpur, Nagpur, Maharashtra
  - Arneja Heart & Multispeciality Hospital, Nagpur, Maharashtra
  - Shri Krishna Hrudayalaya & Critical Care Centre, Nagpur, Maharashtra
  - Sengupta Hospital and Research Institute, Nagpur, Maharashtra
  - B J Goverment Medical College and Sassoon General Hospital, Pune, Maharashtra
  - Jehangir Clinical Development Centre, Pune, Maharashtra
  - Sahyadri Clinical Research And Development Center, Pune, Maharashtra
  - KEM Hospital, Pune, Maharashtra
  - G B Pant Institute of Postgraduate Medical Education and Research, New Delhi, National Capital Territory of Delhi
  - Fortis Escorts Heart Institute, New Delhi, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - VMMC & Safdarjung Hospital, New Dehli, New Delhi
  - Post Graduate Institute of Medical Education & Research_Chandigarh, Chandigarh, Punjab
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - Deep Hospital, Ludhiana, Punjab
  - Fortis Hospital, Mohali, Mohali, Punjab
  - S.P. Medical College and A.G. Hospitals, Bikaner, Rajasthan
  - SMS Medical College & Attached Hospitals, Jaipur, Rajasthan
  - All India Institute of Medical Sciences (AIIMS), Jodhpur, Jodhpur, Rajasthan
  - All India Institute of Medical Sciences (AIIMS), Jodhpur, Rajasthan
  - The Madras Medical Mission, Chennai, Tamil Nadu
  - Osmania General Hospital, Hyderabad, Telangana
  - Guru Nanak CARE Hospitals, Hyderabad, Telangana
  - AIG Hospitals,Hyderabad, Hyderabad, Telangana
  - King George's Medical University (KGMU), Lucknow, Uttar Pradesh
  - Shri Mahant Indiresh Hospital, Dehradun, Uttarakhand
  - IPGME&R and SSKM Hospital, Kolkata, West Bengal
  - Aligarh Muslim University, Aligarh
  - MS Ramaiah, Bengaluru
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre, Karnataka
  - Dr B L Kapur Memorial Hospital, New Delhi
  - Sir Ganga Ram Hospital-Cardiology, New Delhi
  - Aakash Healthcare Super Speciality Hospital, New Delhi
  - Lakshmi Hospital, Palakkad
  - JIPMER, Puducherry
- Ireland (7):
  - St James's CRF, Dublin, Leinster
  - Cork University Hospital, Cork
  - The Heartbeat Trust, Dublin
  - Mater Miscericordiae Hospital, Dublin
  - Mater Private Network - Dublin, Dublin
  - St James's CRF, Dublin
  - Mater Private Network Cork, Mahon, Cork
- Israel (8):
  - Shamir MC - Cardiology Department, Beer Yaakov
  - Hillel Yafe MC - Cardiology Department, Hadera
  - Rambam MC - Heart Failure Unit, Haifa
  - Hadassah Ein Karam MC - Cardio Department, Jerusalem
  - Rabin MC Beilinson - Heart Failure Unit, Petah Tikva
  - Kaplan MC - Heart Failure Unit, Rehovot
  - Sourasky MC - Cardio Vascular Research Center, Tel Aviv
  - Sheba MC - Cardiology Clinical Research Unit, Tel Litwinsky
- Italy (31):
  - ASL Al Di Alessandria - Ospedale Santo Spirito - Casale Monferrato - Cardiologia, Casale Monferrato, Al
  - Ospedale Santo Spirito, Casale Monferrato, Al
  - ASST Papa Giovanni XXIII, Bergamo, Bg
  - AORN "San Pio"- Benevento - UOC Cardiologia Interventistica ed UTIC, Benevento, Bn
  - AORN "San Pio"- Benevento, Benevento, Bn
  - Spedali Civili Brescia, Brescia, Bs
  - AORN "Sant'Anna e San Sebastiano", Caserta, Ce
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro, Cz
  - A.O.U. Ferrara, Sant'Anna, Cona (Ferrara), Fe
  - IRCCS Ospedale Policlinico San Martino, Genova, Ge
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo, Lombardy
  - Azienda Ospedaliera di Perugia;Ospedale S. Maria della Misericordia, Perugia, Pg
  - Fondazione Toscana Gabriele Monasterio - Dipartimento Cardiotoracico - UOC Cardiologia e Medicina Cardiovascolare, Pisa, Pi
  - Fondazione CNR-Regione Toscana Gabriele Monasterio, Pisa, Pi
  - Azienda Sanitaria Locale Roma 1 - Ospedale San Filippo Neri - Cardiologia Clinica, Roma, Rm
  - Azienda Ospedaliera Universitaria Senese, Siena, Si
  - Presidio Ospedaliero di Rivoli, Rivoli, To
  - Azienda Sanitaria Ospedaliera Ordine Mauriziano SC Cardiologia, Torino, To
  - Ospedale Ca' Foncello, Treviso, Veneto
  - AOUI Verona, Verona, Vr
  - Fondazione Salvatore Maugeri I.R.C.C.S. - Bari, Bari
  - Ospedali riuniti di Foggia, Foggia
  - AUSL Toscana Sud Est - Ospedale Misericordia Grosseto, Grosseto
  - ASST Fatebenefratelli Ospedale Luigi Sacco Medicina Interna, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Azienda Ospedaliera Dei Colli - Monaldi - Centro ricerche cardiologiche, Napoli
  - Azienda Ospedaliera di Rilievo Nazionale AORN Dei Colli, "V.Monaldi",, Napoli
  - AOU Maggiore della Carità di Novara - Dipartimento Toraco-Cardio-Vascolare - SCDU Cardiologia, Novara
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Sanitaria Univ Giuliano Isontina - SC Cardiologia, Trieste
  - Azienda Sanitaria Univ Giuliano Isontina, Trieste
- Japan (53):
  - Uwajima City Hospital_Cardiology, Uwajima-shi, Ehime
  - Showa University Fujigaoka Hospital_Cardiology, Yokohama, Kanagawa
  - The Univ. of Tokyo Hp., Dept. of Cardiovascular Medicine, Bunkyo-ku, Tokyo
  - Hamanomachi Hospital_Cardiovascular medicine, Fukuoka
  - Kyushu University Hospital_Cardiovascular Medicine, Fukuoka
  - Fukuoka University Hospital_Cardiology, Fukuoka-shi, Fukuoka
  - Ogaki Municipal Hospital_Cardiology, Gifu
  - JA Shizuoka Kohseiren Enshu Hospital_ Cardiology, Hamamatsu-shi, Shizuoka
  - Hyogo Prefectural HarimaHimeji General Medical Center_Cardiology, Himeji-shi, Hyogo
  - Asahikawa-Kosei General Hospital_Cardiology, Hokkaido
  - Veritas Hospital_Cardiology, Hyōgo
  - National Hospital Organization Mito Medical Center_Cardiovascular medicine, Ibaraki
  - Saiseikai Imabari Hospital_Cardiology, Imabari-shi, Ehime
  - Saiseikai Imabari Hospital, Imabari-shi, Ehime
  - Ishikawa Prefectural Central Hospital_Cardiology, Ishikawa
  - Mitoyo General Hospital_Cardiovascular medicine, Kagawa
  - Kagoshima City Hospital_Cardiovascular Medicine, Kagoshima
  - Yokohama Minami Kyousai Hospital_Cardiology, Kanagawa
  - Kanagawa Prefectural Hospital Organization Kanagawa Cardiovascular and Respiratory Center_Cardiology, Kanagawa
  - Tokai University Hospital_Cardiology, Kanagawa
  - Kishiwada Tokushukai Hospital_Cardiology, Kishiwada-shi, Osaka
  - Japan Community Health care Organization Kyushu Hospital_Cardiology, Kitakyushu-shi, Fukuoka
  - JCHO Kyushu Hospital_Cardiology, Kitakyushu-shi, Fukuoka
  - Rakuwakai Marutamachi Hospital_Cardiology, Kyoto
  - Kyoto University Hospital_Cardiovascular Medicine, Kyoto
  - Mie Prefectural General Medical Center_Cardiology, Mie
  - KKR Tohoku Kosai Hospital_Cardiology, Miyagi
  - Tohoku Medical and Pharmaceutical University Hospital_Division of Cardiology, Miyagi
  - National Hospital Organization Sendai Medical Center_Cardiovascular medicine, Miyagi
  - Iwate Prefectural Central Hospital_Cardiology, Morioka-shi, Iwate
  - Iwate Prefectural Central Hospital, Morioka-shi, Iwate
  - Nagasaki Harbor Medical Center_Cardiovascular medicine, Nagasaki
  - Okayama City General Medical Center Okayama City Hospital_Cardiovascular Medicine, Okayama
  - Okayama Medical Center_Cardiology, Okayama
  - Okayama University Hospital_Cardiovascular Medicine, Okayama-shi, Okayama
  - National Hospital Organization Osaka National Hospital_Cardiovascular Division, Osaka
  - Saiseikai Suita Hospital_Cardiovascular Medicine, Osaka
  - National Cerebral and Cardiovascular Center Hospital_Department of Heart Failure, Osaka
  - Osaka University Hospital_Cardiovascular medicine, Osaka
  - The University of Osaka Hospital_Cardiovascular medicine, Osaka
  - Yao Tokushukai General Hospital_Cardiovascular division, Osaka
  - Saga-ken Medical Centre Koseikan_Cardiology, Saga
  - Chutoen General Medical Center_Cardiology, Shizuoka
  - Kagawa Prefectural Central Hospital_Cardiovascular Medicine, Takamatsu-shi, Kagawa
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Juntendo University Hospital_Cardiology, Tokyo
  - Tokyo Shinagawa Hospital_Cardiovascular Medicine, Tokyo
  - Keio University Hospital_Cardiology, Tokyo
  - Tottori University Hospital_Cardiovascular Medicine, Tottori
  - Toyama University Hospital_Internal Medicine 2, Toyama
  - National Hospital Organization Iwakuni Clinical Center_Cardiovascular Medicine, Yamaguchi
  - JCHO Tokuyama Community Health Center_Department of Cardiology, Yamaguchi
  - Saiseikai Yokohamashi Nanbu Hospital_Cardiology, Yokohama-shi, Kanagawa
- Latvia (9):
  - Zane Lucane GP Practice, Grobiņa, South Kurzeme Municipality
  - Zemgales diabetes centre, Jelgava
  - Riga 1st Hospital, Riga
  - P. Stradins Clinical University Hospital, Riga
  - Adoria, Riga
  - Professor Skride Heart Clinic, Riga
  - GK Neiroklinika, Riga
  - Veselibas centru apvieniba, Riga
  - Riga East Clinical University Hospital - Clinic "Gailezers", Riga
- Lithuania (9):
  - Kaunas Hospital of the Lithuanian University of Health Sciences, Kaunas
  - Klinikiniai sprendimai, Kaunas, Kaunas
  - JSC "Saules seimos medicinos centras", Kaunas
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - Cardiology and Rehabilitation Clinic, Klaipėda
  - Klaipeda university hospital, Klaipėda
  - Republican Siauliai Hospital Consulting Outpatient Clinic, Šiauliai
  - JSC Inlita Santaros, Vilnius
  - Vilnius University hospital Santaros klinikos, Vilnius
- Malaysia (12):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur
  - Hospital Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Sarawak Heart Centre, Kota Samarahan, Sarawak
  - Hospital Serdang, Kajang, Selangor
  - Universiti Teknologi MARA, Sungai Buloh Campus, Sungai Buloh, Selangor
  - Hospital Serdang, Kajang
  - Hospital Kuala Lumpur, Kuala Lumpur
- Mexico (16):
  - Hospital Cardiológica Aguascalientes, Aguascalientes, Aguascalientes
  - CINCAME, Tijuana, Estado de Baja California
  - Diseño y Planeacion en Investigacion Medica S.C., Guadalajara, Jalisco
  - Diseño y Planeación en Investigación Médica S.C., Guadalajara, Jalisco
  - Instituto Nacional de Cardiología Ignacio Chavez, Mexico City, México, D.F.
  - Internal Medicine Clin Trials, Monterrey, Nuevo León
  - Cardiolink Clin Trials S.C., Monterrey, Nuevo León
  - Eukarya Pharmasite S.C., Monterrey, Nuevo León
  - Centro de Investigación y Control Metabólico S. C., San Nicolás de los Garza, Nuevo León
  - Centro de Estudios Clinicos de Querétaro S.C., Santiago de Querétaro, Qro., Querétaro
  - Centro de atención e investigación cardiovascular del Potosí, San Luis Potosí City, San Luis Potosí
  - Centro para el Desarrollo de la Medicina y de Asistencia Médica Especializada, S.C., Culiacán, Sinaloa
  - Centro para el Desarrollo de la Medicina y la Asistencia, Culiacán, Sinaloa
  - Hospital Angeles de Xalapa, Xalapa, Veracruz
  - Centro de Investigación Biomédica y Farmacéutica S.C., Mexico City
  - Centro de Imagen y Tecnologia en Intervención Cardiovascular, México
- Netherlands (11):
  - OLVG Oost, Amsterdam
  - Deventer Ziekenhuis - Cardiologie, Deventer
  - Albert Schweitzer Ziekenhuis locatie Dordwijk, Dordrecht
  - Treant zorggroep, Emmen
  - Medisch Spectrum Twente, Enschede
  - UMC Groningen - Cardiologie, Groningen
  - Zuyderland ziekenhuis - Cardiologie, Heerlen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - Haga Ziekenhuis, The Hague
- North Macedonia (3):
  - PHI City General Hospital 8th September, Skopje
  - PHI University Clinic for Cardiology, Skopje
  - Private Healthcare Institution - Acibadem Sistina Hospital Skopje, Skopje
- Norway (6):
  - Haukeland Universitetssykehus, Bergen
  - Akershus universitetssykehus HF, Lørenskog
  - Colosseumklinikken Medisinske Senter AS, Oslo
  - Rikshospitalet - Kardiologisk forskning, Oslo
  - Oslo universitetssykehus HF - Ullevål, Oslo
  - Stavanger Universitetssykehus, Helse Stavanger HF, Stavanger
- Poland (50):
  - Wojewodzki Szpital Zespolony Im.L.Rydygiera W Toruniu, Torun, Kuyavian-Pomeranian Voivodeship
  - Kardio Life - Tomasz Borkowski, Włocławek, Kuyavian-Pomeranian Voivodeship
  - American Heart of Poland S.A., Chrzanów, Lesser Poland Voivodeship
  - MediNess Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. J.Mikulicza-Radeckiego, Wroclaw, Lower Silesian Voivodeship
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika Samodzielny Publiczny Zaklad Opieki Zdrowotnej We Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Zdrowie S.C. Agnieszka I Donald Drozdz, Wroclaw, Lower Silesian Voivodeship
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni Im.Sw.Jana Pawla II, Grodzisk Mazowiecki, Masovian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Im. Prof. W. Orlowskiego Centrum Medycznego Ksztalcenia Podyplomowego, Warsaw, Masovian Voivodeship
  - Panek Med Centrum Leczenia Chorob Naczyn, Bialystok, Podlaskie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku K. Kardio, Bialystok, Podlaskie Voivodeship
  - Ind. Prak. Lek. w dziedz. Kardiologii lek. med. K. Cymerman, Gdynia, Pomeranian Voivodeship
  - American Heart of Poland S.A., Dąbrowa Górnicza, Silesian Voivodeship
  - Gornoslaskie Centrum Medyczne Im Prof. Leszka Gieca Sląskiego Uniwersytetu Medycznego W Katowicach, Katowice, Silesian Voivodeship
  - Pro Familia Altera Sp. z o.o., Katowice, Silesian Voivodeship
  - Poradnia Aka-Med Centrum Sp. z o.o., Ruda Śląska, Silesian Voivodeship
  - American Heart of Poland S.A., Tychy, Silesian Voivodeship
  - Slaskie Centrum Chorob Serca W Zabrzu, Zabrze, Silesian Voivodeship
  - American Heart of Poland S.A., Bełchatów
  - Szpital Miejski w Gliwicach Sp. z o.o., Gliwice
  - Kardio Brynow Sp. z o. o., Katowice
  - Care Clinic Sp. z o. o., Katowice
  - Gyncentrum Sp. z o. o., Katowice
  - Vita Longa Sp. z o. o., Katowice
  - SCANMED Spółka Akcyjna, Kluczbork
  - Specjalistyczna Praktyka Lekarska L. Bryniarski, Krakow
  - UniCardia & UniMedica & UniEstetica, Krakow
  - Intercard Spolka z ograniczona odpowiedzialnoscia, Krosno
  - Santa Sp. z o.o., Lodz
  - Wojewódzki Specjalistyczny Szpital im.Wl. Bieganskiego,, Lodz
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Clinical Best Solutions Sp. z o.o., Sp. k, Lublin
  - Szpital Sw. Anny w Miechowie, Miechów
  - Jantar Sp. z o.o., Ostrów Wielkopolski
  - Wojewodzki Szpital Im. Sw.Ojca Pio W Przemyslu, Przemyśl
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Ministerstwa Spraw Wewnetrznych i Administracji w Rzeszowie, Rzeszów
  - EMED Centrum Usług Medycznych Ewa Smialek, Rzeszów
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
  - American Heart of Poland S.A., Sztum
  - Balticmed Świnoujście Sp. z o. o., Świnoujście
  - American Heart of Poland S.A., Tychy
  - Polimedica Centrum Badan, Profilaktyki i Leczenia Sp. z o. o., Warsaw
  - Polimedica Centrum Badań, Profilaktyki i Leczenia Sp. z o. o., Warsaw
  - Wojskowy Instytut Medyczny Panstwowy Instytut Badawczy, Warsaw
  - Medical Network Sp. z o. o., Warsaw
  - NZOZ Centrum Medyczne SERAFIN-MED Halina Serafin, Żarów
  - Szpitale Powiatowe Sp. z o.o., Łask
  - American Heart of Poland S.A., Bełchatów, Łódź Voivodeship
  - Uniwersytecki Szpital Kliniczny nr 2 Uniwersytetu Medycznego w Łodzi, Lodz, Łódź Voivodeship
  - American Heart of Poland S.A., Zgierz, Łódź Voivodeship
- Portugal (16):
  - Hospital de Cascais, Alcabideche
  - ULS De Braga, E.P.E. - Hospital de Braga, Braga
  - ULS Do Baixo Mondego, E.P.E. - Hospital Distrital Figueira Da Foz, Figueira da Foz Municipality
  - ULS Da Guarda E.P.E. - Hospital Sousa Martins, Guarda
  - ULS De Tâmega e Sousa E.P.E. - Hospital Padre Américo, Guilhufe - Penafiel
  - ULS Regiao De Leiria E.P.E.- Hospital de Santo André, Leiria
  - Unidade Local De Saude De Lisboa Ocidental E.P.E. - Hospital São Francisco Xavier, Lisbon
  - Hospital Da Luz S.A., Lisbon
  - Hospital da Luz, Lisbon
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Unidade Local De Saude De Santa Maria E.P.E., Lisbon
  - Hospital Cuf Descobertas S.A., Lisbon
  - Unidade Local de Saúde de Santo António, E.P.E, Porto
  - ULS Entre Douro e Vouga E.P.E. - Hospital São Sebastião, Santa Maria da Feira
  - Hospital da Luz Setúbal, Setúbal
  - ULS Da Arrábida, E.P.E._Hospital de São Bernardo, Setúbal
- Romania (34):
  - CMI Dr. Cristian Podoleanu, Târgu Mureş, Targu Mures
  - Cabinet Medical de Cardiologie Dr. Calin Pop, Baia Mare
  - S.C. Centrul Medical Unirea S.R.L., Brasov
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed, Brasov
  - Spitalul Clinic Judetean De Urgenta Brasov, Brasov
  - Spitalul Județean de Urgență Brăila, Brăila
  - "Carol Davila" Military Emergency Hospital, Bucharest
  - Hightech Medical Services S.R.L., Bucharest
  - Spitalul Universitar de Urgență Elias, Bucharest
  - Lotus Med SRL, Bucharest
  - Centrul Medical Emerald, Bucharest
  - Donna Medplus S.R.L., Bucharest
  - Ecocard Srl, Bucharest
  - Davius Clinicmed Srl, Bucharest
  - Institutul De Urgenta Pentru Boli Cardiovasculare Prof. Dr. C. C. Iliescu, Bucharest
  - Spitalul Clinic de Urgenta "Sf. Ioan" Bucuresti, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Mat Cord Biomedica S.R.L., Buzău
  - Spitalul Clinic Judetean De Urgenta Sfantul Apostol Andrei Constanta, Constanța
  - Neurocord Medical SRL, Craiova
  - Cardiomed SRL, Craiova
  - SC Diamed Obesity SRL, Galati
  - Institutul de Boli Cardiovasculare "Prof. Dr. George I.M. Georgescu", Iași
  - SC Consultmed SRL, Iași
  - SC Cardiomed SRL, Iași
  - Spitalul Clinic Judetean De Urgenta Bihor, Oradea
  - Bella Praxis S.R.L., Paşcani
  - Sc Sal Med Srl, Piteşti
  - Spital Judetean De Urgenta Satu Mare, Satu Mare
  - Emergency Institute For Cardiovascular Diseases And Transplant, Târgu Mureş
  - Spitalul Clinic Judetean De Urgenta Targu Mures, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
  - Institutul de Boli Cardiovasculare Timisoara, Timișoara
  - Echipa Medical.33 S.R.L, Timișoara
- Serbia (12):
  - Clinical centre of Serbia, Clinic for cardiology, Belgrade
  - Clinical Centre of Serbia, Emergency Centre, Department of Cardiology, Belgrade
  - Emergency Internal Medicine Clinic, Belgrade
  - General Hospital "Euromedik 2", Belgrade
  - Institute for Cardiovascular Diseases ''Dedinje'', Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Institute for Cardiovascular Diseases of Vojvodina - Sremska Kamenica, Kamenitz
  - University Clinical Centre Kragujevac, Kragujevac
  - Medical center Leskovac, Leskovac
  - University Clinical Centre Nis, Clinic for Cardiology, Niš
  - Medical center Uzice, Užice
- Singapore (6):
  - National University Hospital Singapore, Singapore
  - National Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore
- Slovakia (11):
  - Nemocnica S Poliklinikou Brezno N.O., Brezno, Banská Bystrica Region
  - Interna SK s.r.o., Svidník, Presov
  - Narodny ustav srdcovych a cievnych chorob, a.s., Bratislava
  - KARDIO-SANUS, spol. s r.o., Bratislava
  - CARDIO D&R, s.r.o., Košice
  - Nemocnicna a.s., Malacky
  - MED-CENTRUM, s.r.o., Martin
  - Intradia s.r.o., Nitra
  - BENIMED, s.r.o., Piešťany
  - Fakultna Nemocnica Trnava, Trnava
  - MEDIVASA, s.r.o., Kardiologicka ambulancia 1, 2, Žilina
- Slovenia (3):
  - General hospital Celje - cardiology, Celje
  - UKC Ljubljana, Cardiology department, Ljubljana
  - UKC Maribor - cardiology, Maribor
- South Africa (25):
  - Excellentis Clinical Trial Consultants, George, Eastern Cape
  - Cardiology Research_Bloemfontein, Bloemfontein, Free State
  - IATROS International, Bloemfontein, Free State
  - Josha Research, Bloemfontein, Free State
  - East Rand Physicians, Benoni, Gauteng
  - Johese Clinical Research, Centurion, Gauteng
  - Wits Bara Clinical Trial Site, Johannesburg, Gauteng
  - Dr Garda Cardiology Practice, Johannesburg, Gauteng
  - WITS Clinical Research, Johannesburg, Gauteng
  - Lenasia Clinical Trial Centre, Lenasia, Gauteng
  - Shop#1 Health Emporium, Midrand, Gauteng
  - RYEXO Clinical Research, Pretoria, Gauteng
  - Dr Mpe's Practice, Pretoria, Gauteng
  - Raslouw Private Hospital, Pretoria, Gauteng
  - Synexus Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Clinical Research Institute of South Africa, KwaDukuza, KwaZulu-Natal
  - KwaPhila Health Solutions, Durban, KwwaZulu Natal
  - Synexus Helderberg Clinical Research Centre, Cape Town, Western Cape
  - Dr Corbett, Cape Town, Western Cape
  - Tread Research (Pty)Ltd, Cape Town, Western Cape
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Cardiac Clinical Research Unit, University of Cape Town, Cape Town, Western Cape
  - Dr Hendrik Snyman's Practice, Mossel Bay, Western Cape
  - Synexus Helderberg Clinical Research Centre, Somerset West, Western Cape
  - Clinical Projects Research, Worcester, Western Cape
- South Korea (19):
  - Bucheon Sejong Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
- Spain (17):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Vithas Sevilla, Castilleja de la Cuesta
  - Hospital Univ. de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario La Luz_Cardiología, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Fundación para la Investigación del Hospital Clínico de Valencia (INCLIVA), Valencia
  - Hospital General de Valencia, Valencia
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Kuang Tien General Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District
- Thailand (21):
  - Thammasat University Hospital, Klong Luang, Pathumthani, Changwat Pathum Thani
  - Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - Chulabhorn hospital_Cardiovascular, Bangkok
  - Chulabhorn hospital, Bangkok
  - Cardio-Vajira, Bangkok
  - Vajira Hospital - Cardio, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Ramathibodi Hospital-Cardiovascular metabolic Center, Bangkok
  - Ramathibodi Hospital_Cardiovascular metabolic Center, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital_Cardiology, Chiang Mai
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Chiang Rai Prachanukroh Hospital, Chiang Rai
  - Srinagarind Hospital, Khon Kaen
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima
  - Thammasat Hospital_Cardiology, Pathum Thani
  - Buddhachinaraj Hospital_Cardiology, Phitsanulok
  - Banphaeo General Hospital, Samutsakhon
  - Songklanagarind Hospital, Songkhla
  - Sunpasitthiprasong Hospital_Pediatrics Department, Ubon Ratchathani
  - Sunpasitthiprasong Hospital, Ubon Ratchathani
- Turkey (Türkiye) (18):
  - Afyonkarahisar Health Sciences University, Afyonkarahisar
  - Afyonkarahisar Sağlık Bilimleri Üniversitesi Sağlık Uygulama Ve Araştırma Merkezi- Kardiyoloji, Afyonkarahisar
  - Hacettepe Üniversitesi Hastanesi- Kardiyoloji, Ankara
  - Ankara Bilkent Şehir Hastanesi-Kardiyoloji, Ankara
  - Ankara Sehir Hastanesi Cardiology, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Akdeniz Üniversitesi Hastanesi-Kardiyoloji, Antalya
  - Trakya Üniversitesi Tıp Fakültesi Hastanesi- Kardiyoloji, Edirne
  - Eskişehir Osmangazi Üniversitesi Hastanesi- Kardiyoloji, Eskişehir
  - İstanbul Üniversitesi-Cerrahpaşa Tıp Fakültesi Kardiyoloji Enstitüsü, Istanbul
  - Mehmet Akif Ersoy Göğüs Kalp ve Damar Cerrahisi EAH, Istanbul
  - Mehmet Akif Ersoy Thoracic and Cardiovascular Surgery Training Research Hospital_Istanbul, Istanbul
  - Dr. Siyami Ersek Göğüs Kalp ve Damar Cerrahisi EAH- Kardiyoloji, Istanbul
  - Ege Üniversitesi Hastanesi- Kardiyoloji, Izmir
  - Dokuz Eylül Üniversitesi Araştırma Uygulama Hastanesi-Kardiyoloji, Izmir
  - Erciyes Üniversitesi Hastanesi- Kardiyoloji, Kayseri
  - Kocaeli Üniversitesi Hastanesi- Kardiyoloji, Kocaeli
  - Mersin Üniversitesi Hastanesi- Kardiyoloji, Mersin
- United Kingdom (22):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Basildon University Hospital, Basildon, Essex
  - University Hospital Monklands - Cardiology Research, Airdrie, Lanarkshire
  - St George's Hospital - Cardiology, Tooting, London
  - St George's Hospital, Tooting, London
  - University Hospital Hairmyres - Cardiology, East Kilbride, South Lanarkshire
  - St. Richard's Hospital_Cardiology, Chichester, West Sussex
  - St. Richards Hospital, Chichester, West Sussex
  - Aberdeen Royal Infirmary, Aberdeen
  - Southmead Hospital, Bristol
  - Craigavon Area Hospital_Cardiovascular Research Unit, Craigavon
  - Royal Bournemouth Hospital, Dorest
  - Royal Devon and Exeter Hospital, Exeter
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Glasgow Royal Infirmary, Glasgow
  - Wycombe General Hospital, High Wycombe
  - Aintree University Hospital, Liverpool
  - Manchester Royal Infirmary - Manchester Heart Centre, Manchester
  - North Tyneside General Hospital, North Shields
  - The Royal Oldham Hospital_Cardiology Outpatients Dept., Oldham
  - John Radcliffe Hospital, Oxford
  - University of North Tees Hospital, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com